CLINICAL TRIAL: NCT01855425
Title: Cone Beam CT (CS 9300) for Diagnosis of Select Otorhinolaryngology (ENT) Indications at Lower Dose
Brief Title: Cone Beam CT for Diagnosis of Select Otorhinolaryngology (ENT) Indications at Lower Dose
Acronym: CBCT-ENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carestream Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6K0377
Record Dates: First submitted 2013-05-06; First posted 2013-05-16 (Estimated); Results first posted 2018-08-01 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: CerebroSpinal Fluid (CSF) Leak; Chronic Otitis Media; Otospongiosis; Otosclerosis; Pulsatile Tinnitus; Cholesteatoma
MeSH Terms: conditions — Otosclerosis; Tinnitus; Cholesteatoma | interventions — Radiation

STUDY DESIGN:
Intervention Model Description: Predicate CT Scan and Investigational Cone Beam Scan
Oversight: Data Monitoring Committee: No

ARMS (1):
- Investigational CBCT (Other): Radiation
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Subjects to receive standard of care CT scan and additional Cone Beam CT scan.

SUMMARY:
The study objective is to compare the CBCT images generated by the CS 9300 to those generated by conventional CT.

DETAILED DESCRIPTION:
The study objective is to compare the CBCT images generated by the CS 9300 to those generated by conventional CT. It proposes a direct comparison of diagnostic image quality between the CS 9300 and CT for the ability to view and confirm ENT disorders.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18-80 years of age
* Subjects has provided informed consent
* Subjects must present with symptoms and/or pathology of the sinus or temporal bone region.
* Subject scheduled for additional radiological follow-up and/or endoscopy/surgery.
* CBCT exam performed within a maximum of 2 days of the conventional CT.

Exclusion Criteria:

* Subjects under the age of 18 years, or over the age of 80 years
* Unable to collect all required case information
* Subjects not willing to consent, or consent is withdrawn
* Women in pregnancy or suspected of being pregnant confirmed by pregnancy test

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2012-09-21 (Actual); Primary Completion 2013-08-09 (Actual); Study Completion 2013-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Reh, MD, Principal Investigator — Johns Hopkins Medical Center
Locations (3):
- Johns Hopkins Medical Center, Baltimore, Maryland, United States
- Sint-Augustinus Hospital, Antwerp, Belgium
- C.H.U Bicetre, Paris, France

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational CBCT: Investigator orders Medical CT as part of Standard of Care. Subject consents to be in study and they are also given a Cone Beam CT.
  Radiation: Subjects to receive standard of care CT scan and additional Cone Beam CT scan.
Period: Overall Study
Arm/Group | Investigational CBCT
Started | 96
Completed | 76
Not Completed | 20
Not completed — Physician Decision | 20

BASELINE CHARACTERISTICS:
Groups:
- Investigational CBCT: Investigator orders CT as part of Standard of Care. Subject consents to be in study and they are also given a Cone Beam CT.
  Radiation: Subjects to receive standard of care CT scan and additional Cone Beam CT scan.
Arm/Group | Investigational CBCT
Number analyzed (Participants) | 96
Age, Customized [Number; unit: participants]
  > 18 years - < 80 years | 96
Sex: Female, Male [Count of Participants; unit: Participants] — gender data was not collected
  Participants
    Female | NA — gender data was not collected
    Male | NA — gender data was not collected
Region of Enrollment [Number; unit: participants]
  Belgium | 32
  United States | 19
  France | 45

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With >=3 Diagnostic Rating Using Radlex Scale
Description: Percentage of Participants with >=3 Diagnostic Rating Using Radlex Scale. Five radiologists participated in reader study using Radlex scale below to analyze and rate participant images. They determined if they could make a medical diagnosis for ENT patients.
  Used Radlex Scale - 1-Non-diagnostic, Unacceptable for diagnostic purposes. 2-Limited Acceptable, with some technical defect. 3-Diagnostic, Image quality that would be expected routinely when imaging cooperative patients. 4-Exemplary, Good most adequate for diagnostic purposes.
Time Frame: 11 months
Population: 96 participants were imaged for this study, but only 76 participant image pairs were analyzed in the reader study. 20 participant image pairs were disqualified by the physicians due movement/unclear image quality.
Measure: Mean (Standard Deviation); unit: percentage of participants
Groups:
- Investigational CBCT: Investigational CBCT images
Arm/Group | Investigational CBCT
Number analyzed (Participants) | 76
percentage of participants | 92.63 (4.9)

ADVERSE EVENTS:
Time Frame: 11 months
Arm/Group | Investigational CBCT
All-Cause Mortality (participants affected / at risk) | 0/96
Serious Adverse Events (participants affected / at risk) | 0/96
Other Adverse Events (participants affected / at risk) | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No